CLINICAL TRIAL: NCT02125318
Title: A Phase 2, Open Label Efficacy and Safety Study of Anagrelide Controlled Release (CR) in Subjects With Thrombocytosis Secondary to Essential Thrombocythemia and Other Myeloproliferative Neoplasms (MPN)
Brief Title: A Study of Anagrelide Controlled Release (GALE-401) in Patients With High Platelet Counts Due to Bone Marrow Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galena Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GALE-401-201
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Thrombocytosis; Myeloproliferative Neoplasms
Keywords: myeloproliferative neoplasm; chronic myelogenous leukemia; polycythemia vera; primary myelofibrosis; essential thrombocythemia; anagrelide; thrombocytosis; GALE-401
MeSH Terms: conditions — Thrombocytosis; Myeloproliferative Disorders; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anagrelide CR (GALE-401) (Experimental)
  Interventions: Drug: Anagrelide CR

INTERVENTIONS:
Drug: Anagrelide CR — Starting dose of 0.5 mg b.i.d. (1.0 mg/day) titrated at weekly intervals, on an individual basis, to achieve the lowest dose required to achieve and maintain a target platelet count of 150 - 400 x 10e9/L, tolerability permitting. The dose will be increased at weekly intervals in steps not exceeding 0.5 mg/day; the rate of dose titration may be reduced (i.e., up to once every 2 weeks) at the discretion of the Investigator.
  Other Names: GALE-401

SUMMARY:
Anagrelide is a drug that has been shown to slow down how fast platelets are made in the bone marrow, and has been approved by the FDA for treating high platelets counts in patients with bone marrow disorders.

Anagrelide Controlled Release ("CR") is a new preparation of anagrelide that is made to dissolve more slowly than currently marketed versions of this drug. Because of this, the anagrelide is taken up into the blood more slowly. Researchers think that this slower release of the drug could help to lower side effects that might be caused by high blood levels when the drug dissolves as quickly as it does with the currently marketed product.

The main purposes of this study are to see how well Anagrelide CR can control platelet counts in patients with high platelet levels, to see what kind of side effects it causes, and to measure blood levels of the drug.

DETAILED DESCRIPTION:
This is an open-label, single-arm, multicenter, Phase 2 study of anagrelide CR in subjects with an MPN-related thrombocytosis. Eligible subjects will include those who have not been previously treated for thrombocytosis or have not received platelet-lowering therapy for at least 2 weeks prior to study treatment. Each subject will receive anagrelide CR at a starting dose of 0.5 mg b.i.d. (1.0 mg/day), and is anticipated to continue study treatment for at least 24 weeks. Subjects who have achieved clinical benefit in the opinion of the Investigator and who are tolerating the study drug may continue study treatment until they develop unacceptable toxicity or other discontinuation criteria have been met.

The primary efficacy endpoint will be the proportion of subjects who achieve a platelet response (CR or PR). The safety and tolerability of study treatment will be assessed by the frequency and severity of adverse events as determined by NCI Common Terminology Criteria for Adverse Events (CTCAE) v 4.03. The PK profile of anagrelide CR will be assessed at the initial (0.5mg b.i.d.) and final titrated dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study specific procedure
2. Male or female patients aged ≥ 18 years
3. Diagnosis of a myeloproliferative neoplasm (i.e., chronic myelogenous leukemia (CML), polycythemia vera (PV), primary myelofibrosis (PMF), essential thrombocythemia (ET)) as determined by the treating physician, such as based on the 2008 World Health Organization (WHO) classification of myeloid malignancies
4. Baseline platelet count ≥600 x 10e9/L as determined on two occasions at least 14 days apart prior to the first dose of study drug
5. Requirement for platelet reduction therapy as assessed by the Investigator
6. Currently not receiving therapy specifically intended to reduce platelet counts
7. For patients with ET, prior platelet lowering therapy (e.g., hydroxyurea, anagrelide or interferon) may not be administered within 2 weeks prior to the first dose of study drug.

   For patients with MPN diagnoses other than ET, concurrent anti-MPN treatment is permitted provided that the treatment has been administered at stable doses for at least 4 weeks prior to the first dose of study drug. Examples of permitted medications include but are not limited to hydroxyurea for PV, ruxolitinib for MF, and imatinib for CML. All patients must have discontinued anagrelide at least 2 weeks prior to the first dose of study drug.

   EXCEPTION: busulfan, melphalan and phosphate P-32 must have been discontinued at least 4 weeks prior to the first dose of study drug.
8. Adequate hepatic function defined as bilirubin ≤1.5 x ULN, INR ≤1.5 x ULN, albumin >3.5 g/dL, ALT < 3.0 x ULN, AST < 3.0 x ULN
9. If female, must be of non-childbearing potential, i.e. post- menopausal (defined as > 12 months since last menstrual period) or surgically sterilized (i.e. tubal ligation or hysterectomy at least 6 months prior to screening) or, if of childbearing potential, must not be pregnant or nursing
10. Males and females of child bearing must agree to use an acceptable form of birth control until 28 days following the last dose of study drug

Exclusion Criteria:

1. Other MPN diagnoses not specifically included above: Chronic neutrophilic leukemia, chronic eosinophilic leukemia, mastocytosis, and unclassifiable MPNs
2. Previously found to be refractory to anagrelide therapy (i.e., failure to achieve a platelet count <600 x 10e9/L for reasons other than anagrelide-related toxicity)
3. History of coronary artery disease requiring a revascularization procedure within 3 months prior to screening
4. Left bundle branch block or sustained ventricular tachycardia (>30 seconds) evident on 12-lead ECG at screening
5. Tachycardia defined as resting heart rate >100 bpm at screening
6. Unstable angina (characterized by increasingly frequent episodes with modest exertion or at rest, worsening severity, or prolonged duration) within 3 months prior to screening
7. Transient ischemic attack (TIA) or stroke within 3 months prior to screening
8. Unstable or clinically significant concurrent medical condition that would, in the opinion of the Investigator, jeopardize the safety of a subject and/or their compliance with the protocol.
9. Current alcohol or drug abuse, or a significant medical condition that, in the opinion of the Investigator, may impair compliance with the requirements of the protocol
10. History of allergic hypersensitivity to anagrelide or any component of its formulations
11. Administration of Type 3 phosphodiesterase (PDE3) inhibitors (e.g., inamrinone, cilostazol, milrinone) within 2 weeks prior to initiating study treatment
12. Administration of any investigational product within 4 weeks prior to initiating study treatment
13. History of intolerance of other PDE3 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Platelet Response | Up to 24 weeks
  The primary efficacy endpoint will be the proportion of subjects who achieve a platelet response (complete or partial response), with response defined according to the following criteria:
  * Complete response (CR): platelet count of ≤400 x 10e9/L maintained for at least 4 weeks
  * Partial response (PR): a platelet count of ≤600 x 10e9/L or a ≥50% reduction from baseline and maintenance of the reduction for at least 4 weeks
  * Nonresponse: failure to meet CR or PR criteria

SECONDARY OUTCOMES:
Number of subjects with adverse events | Throughout study treatment (expected average of 12 months)
  Frequency and severity of adverse events as determined by NCI CTCAE (v 4.03).
Plasma concentrations of anagrelide | Up to 13 weeks
  Monitor anagrelide levels during dose titration and assess pharmacokinetic profile at starting and final dose levels.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - East Valley Hematology and Oncology Medical Group, Burbank, California
  - California Cancer Associates for Research & Excellence (cCARE), Encinitas, California
  - California Cancer Associates for Research & Excellence (cCARE), Escondido, California
  - California Cancer Associates For Research and Excellence, Fresno, California
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Gettysburg Cancer Center, Hillsdale, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, New Braunfels, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas